CLINICAL TRIAL: NCT06398340
Title: Identifying Physiological Biomarkers for Monitoring Dietary Behaviours
Brief Title: Identifying Wearable Biomarkers to Monitor Dietary Intake
Acronym: FoodSense
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 23HH8489
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Energy Intake; Metabolism; Digestion; Wearables; Dietary Intake Assessment; Healthy Volunteers; Blood Glucose
Keywords: Dietary intake monitoring; wearable sensors; digital health; blood glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Calorie, Then Low Calorie (Experimental): Subjects will receive an unhealthy meal that against the healthy eating guidelines. After a washout period of at least 24hours, subjects will receive a balanced diet that meets healthy eating guidelines.
  Interventions: Other: High Calorie Meal Intervention; Other: Low Calorie Meal Intervention
- Low Calorie, Then High Calorie (Experimental): Subjects will receive a balanced diet that meets healthy eating guidelines. After a washout period of at least 24hours, subjects will receive an unhealthy meal that against the healthy eating guidelines
  Interventions: Other: High Calorie Meal Intervention; Other: Low Calorie Meal Intervention

INTERVENTIONS:
Other: High Calorie Meal Intervention — Subjects will receive a unhealthy meal high in calorie, sugar and fat
Other: Low Calorie Meal Intervention — Subjects will receive a healthy meal with balanced macronutrient, high in vegetables and dietary fibre

SUMMARY:
Background: Measuring what people eat is a challenge in nutrition research. Traditional methods, like food diaries, rely on self-reporting of individuals, and suffer from poor accuracy and recall bias.

Aims: This project aims to identify physiological biomarkers related to food and energy intake, which may be used to develop an objective tool to estimate individuals' food intake in future. Eating behaviours are accompanied by significant physiological changes such as skin temperature, blood oxygen saturation, pulse rate etc. The investigators intend to investigate whether monitoring these physiological changes can help us estimate eating behaviour, such as meal size, eating speed, and duration of meals.

Study design: Ten healthy adults will be invited for two study visits at NIHR Imperial Clinical Research Facility. Each visit will last for approximately 2 hr. They will consume a high- and low-calorie meal designed by nutritional researchers in a randomised order. During eating events, the investigators will track their physiological changes via a bedside monitor and wearable sensors. Blood samples will be taken from participants to measure their glycaemic response. Associations between energy load, glycaemic response, and physiological changes will be investigated. Our findings may promote an accelerated development of a wearable tool for dietary assessment in future.

DETAILED DESCRIPTION:
1 Participants

10 healthy male and female participants. This is a pilot study in a new area and therefore a formal power calculation is not possible.

2. Recruitment

Participants will be recruited from existing healthy volunteer databases and by advertisement in public places. Adverts may be placed in newspapers and put up in public buildings. A contact number on the advert will enable potential participants to contact the research team at Imperial College London. Participation in the study will be entirely voluntary. No undue influence will be exerted by the researchers. Participants will be free to withdraw from the study at any time.

3 Pre-Screening Questionnaire

A pre-screening questionnaire considering the inclusion and exclusion criteria will be completed to establish eligibility. For subjects who complete the questionnaire but do not continue to participate, their data will not be saved.

4 Informed Consent

All participants will sign informed consent before starting the study (at the beginning of the 1st main study visit).

5 Main Study Visits

Ten healthy subjects will attend two study visits at National Institute for Health and Care Research (NIHR) Imperial College London Clinical Research Facility (post code: W12 0NN, London, UK). The participants will consume a high- and low-calorie meal designed by nutritional researchers, in a randomised order. Randomization will be performed using the sealed envelope website by an independent researcher (i.e., not linked to the study). During eating events, physiological changes such as skin temperature, blood oxygen saturation, pulse rate etc and eating movements will be measured via a bedside monitor and non-invasive, wearable sensors. Blood samples will be taken at pre-determined time-points, starting 5 minutes before the meal and lasting for 60 minutes postprandially (at -5, +15, +30, +45, +60 min ). A total of 25 ml blood will be taken per visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18-65 years (inclusive)
* Body mass index (BMI) of 18-30 kg/m2
* Willingness and ability to give written informed consent.
* Willingness and ability to understand, to participate and to comply with the study requirements

Exclusion Criteria:

* Outside of specified age and BMI range
* Chronic medical conditions including for eating disorders, diabetes, obesity, hypertension, cancer, acute infectious disease, renal disease, cardiovascular disease, and chronic gastrointestinal condition.
* Taking part in another research study or donating any blood in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes of heart rate associated with dietary events (pre- vs post- meal). | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Heart rate in bpm before, during and after the dietary event
Changes of blood pressure associated with dietary events (pre- vs post- meal). | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Systolic and diastolic blood pressure in mmHg before, during and after the dietary event
Changes of oxygen saturation associated with dietary events (pre- vs post- meal). | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Oxygen saturation in % before, during and after the dietary event
Changes of skin temperature associated with dietary events (pre- vs post- meal). | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Skin temperature in celsius before, during and after the dietary event
Changes of hand movements associated with dietary events (pre- vs post- meal). | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Hand movements recorded in sensors before, during and after the dietary event

SECONDARY OUTCOMES:
Changes of heart rate associated with energy intake (high vs. low calorie meals) | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Differences on heart rate in bmp between high and low calorie meals
Changes of blood pressure associated with energy intake (high vs. low calorie meals) | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Differences on systolic and diastolic blood pressure in mmHg between high and low calorie meals
Changes of heart oxygen saturation associated with energy intake (high vs. low calorie meals) | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Differences on systolic and diastolic blood pressure in mmHg between high and low calorie meals
Changes of skin temperature associated with energy intake (high vs. low calorie meals) | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Differences on skin temperature in celsius between high and low calorie meals
Changes of hand movements associated with energy intake (high vs. low calorie meals) | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Hand movements recorded in sensors between high and low calorie meals
Vital signs associated with blood glucose, insulin and hormonal levels | Starting 5 minutes before the meal and lasting for 60 minutes postprandially.
  Correlation (expressed in correlation coefficient R) between vital signs (i.e., heart rate in bpm, blood pressure in mmHg, oxygen saturation in %, and skin temperature in celsius )and the blood glucose (mmol/L), insulin (mmol/L)and GIP (mmol/L) response in 60min (reported in area under curve mmol/L*min）

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhu Cai, PhD, Study Chair — Nutrition Research Section, Imperial College London; Mayue Shi, PhD, Principal Investigator — Department of Electrical and Electronic Engineering, Imperial College London
Locations (1):
- NIHR Imperial College London Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi M, Zhou J, Cai M. Multiple physiological and behavioural parameters identification for dietary monitoring using wearable sensors: a study protocol. BMC Nutr. 2025 Oct 6;11(1):183. doi: 10.1186/s40795-025-01168-1. PMID 41053911

DOCUMENTS (2):
  • Study Protocol (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT06398340/Prot_000.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT06398340/ICF_001.pdf